CLINICAL TRIAL: NCT07098871
Title: The Role of Preoperative Rectus Abdominis and Diaphragm Muscle Thickness in Predicting Postoperative Complications in Patients Undergoing Surgery for Gastrointestinal Malignancies: A Prospective Observational Study
Brief Title: Predictive Value of Preoperative Rectus and Diaphragm Muscle Thickness for Postoperative Complications in Gastrointestinal Cancer Surgery
Status: Recruiting | Type: Observational
Sponsor: Ankara Oncology Research and Training Hospital (Network)
Responsible Party: Principal Investigator, Burak Dincer, Principal Investigator, Ankara Oncology Research and Training Hospital
Other Study IDs: 2025-03/50
Record Dates: First submitted 2025-06-22; First posted 2025-08-01 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Gastrointestinal Cancers; Complication
Keywords: Gastrointestinal Cancers; Postoperative Complications; Rectus Muscle Thickness; Diaphragma Muscle Thickness
MeSH Terms: conditions — Gastrointestinal Neoplasms; Postoperative Complications | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surgery: Patients undergone surgery for gastrointestinal system malignancies
  Interventions: Diagnostic Test: Ultrasonography (Rectus and diaphragma muscle thickness measurement)

INTERVENTIONS:
Diagnostic Test: Ultrasonography (Rectus and diaphragma muscle thickness measurement) — Rectus and diaphragma muscle thickness will be measured by ultrasonography preoperatively.

SUMMARY:
The aim of this observational study is to investigate the relationship between preoperative rectus abdominis and diaphragm muscle thickness and postoperative complication rates in patients undergoing surgery for gastrointestinal system malignancies.

The main research question is whether rectus abdominis and diaphragm muscle thickness can be used to predict postoperative complications in these patients, and whether there are specific cut-off values for these muscle thicknesses.

Participants will be selected from operable gastrointestinal malignancy cases, and preoperative measurements of rectus abdominis and diaphragm muscle thickness will be performed using ultrasonography.

DETAILED DESCRIPTION:
Background and Aim:

Gastrointestinal system (GIS) malignancies are commonly encountered and carry a significant risk of serious complications following surgery. Therefore, several studies in the literature have focused on identifying parameters that can predict the risk of postoperative complications in patients undergoing surgery for GIS malignancies. Some publications have suggested that preoperative nutritional indices may help predict the development of complications, evaluating specific parameters through biochemical tests or radiological assessments of muscle and fat mass.

In our study, we aim to investigate the relationship between preoperative rectus abdominis and diaphragm muscle thickness-measured via ultrasonography during routine fascial block procedures-and the rate of complications occurring within the first 30 days postoperatively in patients undergoing surgery for GIS malignancies.

Methodology:

Patients whose rectus abdominis and diaphragm muscle thickness were measured during routine preoperative fascial block ultrasonography will be included in the study. No additional intervention or procedure is planned; patients will be evaluated as part of standard clinical practice, and their postoperative outcomes will be recorded observationally. No additional tests requiring reimbursement from the national health insurance system will be performed as part of the study.

Study Hypotheses:

H₀ (Null Hypothesis): There is no significant difference in rectus abdominis and diaphragm muscle thickness between patients who develop complications within the first 30 days after GIS malignancy surgery and those who do not.

H₁ (Alternative Hypothesis): There is a significant difference in rectus abdominis and diaphragm muscle thickness between patients who develop complications within the first 30 days after GIS malignancy surgery and those who do not.

Data Collection Tools:

Data will be collected prospectively from routine clinical evaluations. Ultrasonographic measurements of rectus abdominis and diaphragm muscle thickness will be performed by the researchers during routine preoperative fascial block procedures. No additional tests or procedures requiring reimbursement from SGK will be performed. Patient identities and personal data will be kept confidential by the researchers, and all procedures carried out within the study will pose no additional risk to the patients.

Statistical Analysis:

Data obtained from the study will be analyzed using SPSS (Statistical Package for the Social Sciences) version 25.0 (IBM Corp., Armonk, NY, USA). Descriptive statistics (e.g., number, percentage, median) will be used to summarize the data. Quantitative variables will be evaluated using the t-test or Mann-Whitney U test, while categorical variables will be analyzed using the chi-square test or Fisher's exact test. The relationship between rectus and diaphragm muscle thickness and the development of complications will be assessed using receiver operating characteristic (ROC) curve analysis. A p-value of <0.05 will be considered statistically significant, and 95% confidence intervals will be reported.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Patients scheduled for laparoscopic or open surgery due to GIS malignancy between 01.05.2025 and 01.11.2025
* Postoperative follow-up at our center for a minimum of 30 days

Exclusion Criteria:

* Age under 18 years
* Patients not undergoing surgery
* Patients undergoing surgery for indications other than GIS malignancy
* Patients with follow-up data shorter than 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with operable gastrointestinal system cancer from tertiary cancer center
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Correlation between rectus muscle thickness and clavien-dindo grade of postoperative complications | From enrollment to 30th postoperative day.
  Correlation between rectus muscle thickness and clavien-dindo grade of postoperative complications
Correlation between diaphragma muscle thickness and clavien-dindo grade of postoperative complications | From enrollment to 30th postoperative day.
  Correlation between diaphragma muscle thickness and clavien-dindo grade of postoperative complications

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Oncology Training and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No